CLINICAL TRIAL: NCT00910260
Title: Impact on UVB Narrow Band and UVA1 Therapy on Serum 25-hydroxyvitamin D Levels
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 0000
Record Dates: First submitted 2009-04-17; First posted 2009-05-29 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Skin Disease
Keywords: vitamin D level under phototherapy
MeSH Terms: conditions — Skin Diseases | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood analysis — Serum 25-hydroxyvitamin D, calcium, parathormone, phosphate, C-reactive protein and albumin levels will be measured at every visit: day 0, day 7 and day 84.

SUMMARY:
We plan to investigate the serum elevation of 25(OH)D under UVB nb and UVA1 therapy, in order to determine the effect of these nowadays frequently used wavelengths for phototherapy on vitamin D plasma levels. We hope for a better understanding of steady-state and treatment-induced levels of vitamin D changes to better recognize the impact of phototherapy on vitamin D synthesis in the skin, the dimension of vitamin D production to be expected in the course of standard phototherapy and a potential gap in vitamin D production compared to physiological needs which then should be supplemented orally.

DETAILED DESCRIPTION:
This is an open observational study in dermatological patients undergoing phototherapy.

In patients with a skin disease and the routinely given indication for a phototherapy with UVB narrow-band (UVB nb, 311nm) or UVA1 (340-400 nm), the serum 25-hydroxyvitamin D, calcium, parathormone, phosphate and albumin levels will be measured before, during and after completion of the 12-week therapy (30 patients per group). Patients will be recruited in the department of dermatology of the University Hospital Zürich in the outpatient clinic. Following oral and written consent, serum 25-hydroxyvitamin D, calcium, parathormone, phosphate and albumin levels will be measured before the therapy, one week after start as well as after completion of the UVB nb/UVA1 therapy.

In parallel to the study the patients will be asked to fill in a questionnaire evaluating the daily vitamin D consume (milk and milk products, fish, food enhanced in vitamin D, multivitamin supplements), sun exposure per week during previous weeks, degree of tanning, the use of sunscreen, the DLQI and Skindex-29.

A physical examination including clinical score where available will be performed at every "checkpoint". During the first physical examination the Fitzpatrick-skin type of patient will be recorded.

The following participant characteristics will be recorded: age, weight, body mass index (BMI), phototype, skin disease, comorbidities, usual medication, and period of the year where UVB nb/UVA1 therapy is performed (summer vs. winter), cumulative UVB nb/UVA1 doses.

ELIGIBILITY:
Inclusion criteria:

1. Dermatological indication for a phototherapy with UVB nb or UVA1
2. Oral and written informed patient consent

Exclusion criteria:

1. Interruption of the light therapy for more than 14 days
2. Withdrawal of consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dermatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Determination of baseline serum 25-hydroxyvitamin D, calcium, parathormone, phosphate and albumin levels before therapy | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Dermatology Department, University Hospital, Zurich, Switzerland